CLINICAL TRIAL: NCT03451487
Title: A Randomized, Single-blind, Parallel Group and Multiple - Dose Design Study to Evaluate the Pharmacokinetics of Acetaminophen and Its Toxic Metabolites With Panadol® and Various Formulations of SafeTynadol® in Healthy Volunteers
Brief Title: A Randomized, Single-blind, Parallel Group and Multiple - Dose Design Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinew Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Oral AAP-001
Record Dates: First submitted 2018-02-24; First posted 2018-03-01 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-04

CONDITIONS: Acetaminophen Toxicity
Keywords: acetaminophen; acute liver failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Single Blindie
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Reference drug (1000mg) (Placebo Comparator): Eligible subjects were randomly assigned to either of the two treatment sequence.The evaluable subjects were those who had completed both period I and II. The study was completed when there were at least 12 evaluable subjects.
  Panadol® oral dosage form (500 mg*2 tablets = 1000 mg) was orally administered with 240 ml of water once daily in the morning in each of the single-dose study period.
  Interventions: Drug: Panadol®
- Test drug (1000mg) (Experimental): Eligible subjects were randomly assigned to either of the two treatment sequence.The evaluable subjects were those who had completed both period I and II. The study was completed when there were at least 12 evaluable subjects.
  SafeTynadol® oral dosage form (500 mg*2 tablets = 1000 mg) was orally administered with 240 ml of water once daily in the morning in each of the single-dose study period.
  Interventions: Drug: SafeTynadol®
- Reference drug (4000mg) (Placebo Comparator): Eligible subjects were randomly assigned to either of the two treatment sequence.The evaluable subjects were those who had completed both period III and IV. The study was completed when there were at least 12 evaluable subjects.
  Panadol® oral dosage form (500 mg*8 tablets = 4000 mg) was orally administered with 240 ml of water once daily in the morning in each of the single-dose study period.
  Interventions: Drug: Panadol®
- Test drug (4000mg) (Experimental): Eligible subjects were randomly assigned to either of the two treatment sequence.The evaluable subjects were those who had completed both period III and IV. The study was completed when there were at least 12 evaluable subjects.
  SafeTynadol® oral dosage form (500 mg*8 tablets = 4000 mg) was orally administered with 240 ml of water once daily in the morning in each of the single-dose study
  Interventions: Drug: SafeTynadol®
- Reference drug 2 tablets Q6H (28,000mg) (Placebo Comparator): Eligible subjects were randomly assigned to either of the two treatment stage.Each treatment will be completed when there are at least 7 evaluable subjects. The evaluable subjects are randomized into period V.
  Panadol® oral dosage form (500mg*2 tablets =1000mg) will be orally administered with 240 ml of water every 6 hours daily in each of the multiple-dose study period (Q6H, total 28 dosages, 56 tablets).
  Interventions: Drug: Panadol®
- Test drug 2 tablets Q6H (28,000mg) (Experimental): Eligible subjects were randomly assigned to either of the two treatment stage.Each treatment will be completed when there are at least 7 evaluable subjects. The evaluable subjects are randomized into period V.
  SafeTynadol® oral dosage form (500mg*2 tablets =1000mg) will be orally administered with 240 ml of water every 6 hours daily in each of the multiple-dose study period (Q6H, total 28 dosages, 56 tablets).
  Interventions: Drug: SafeTynadol®

INTERVENTIONS:
Drug: Panadol® — Acetaminophen 500mg Tablet
  Other Names: Acetaminophen
  Arms: Reference drug (1000mg); Reference drug (4000mg); Reference drug 2 tablets Q6H (28,000mg)
Drug: SafeTynadol® — Acetaminophen 500mg Tablet
  Other Names: SNP-810
  Arms: Test drug (1000mg); Test drug (4000mg); Test drug 2 tablets Q6H (28,000mg)

SUMMARY:
To investigate and compare the possible response of Panadol® and SafeTynadol® formulations in healthy volunteers.

DETAILED DESCRIPTION:
Acetaminophen (AAP) is the most popular used analgesic/ antipyretic drug with serious hepatotoxic adverse effects; suicidal or unintentional overdose of AAP-induced hepatotoxicity. Cytochrome P450 2E1 (CYP2E1) is thought contribute to the responsible reactive metabolite N-acetyl-p-benzoquinone (NAPQI) of AAP overdose-induced hepatotoxicity. Pharmaceutical excipients are inactive ingredients that are added to a pharmaceutical compound. The objective of this study was to investigate the possible response of Panadol® (AAP alone) and SafeTynadol® (AAP with various selected excipients combination) formulations, while observing the AAP toxic metabolites (AAP-Cys) circumstances change in healthy volunteers. According to the current safety data, could be potentially develop hepatotoxicity-free AAP new formulation drug.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy adult subjects between 20-50 years of age.
2. Body weight within 80-120% of ideal body weight. Male: Ideal body weight = (height - 80) * 0.7 Female: Ideal body weight = (height - 70) * 0.6
3. Acceptable medical history and physical examination including:

   * normal ECG results within six months prior to Period I (or Period III or Period V) dosing.
   * no particular clinical significance in general disease history within two months prior to Period I (or Period III or Period V) dosing.
4. Acceptable clinical laboratory determinations without significant deviation from normal values within two months prior to Period I (or Period III or Period V) dosing, which includes AST (SGOT), ALT (SGPT), r-GT, alkaline phosphatase, total bilirubin, albumin, glucose, BUN, uric acid, creatinine, total cholesterol, triglyceride (TG) and oral galactose single point (OGSP).
5. Acceptable hematology within two months prior to the study, which includes hemoglobin, hematocrit, red blood cells, MCV, MCH, MCHC, white blood cells, differential white blood cells and platelets.
6. Acceptable urinalysis within two months prior to the study, which includes pH, blood, glucose and protein.
7. Signed the written informed consent to participate in this study.

Exclusion Criteria:

1. History or presence of alcohol abuse, defined as consumption of more than 210 mL of alcohol per week (the equivalent of 14 glasses of 120-mL wine or 14 cans of 350-mL beer), or other substance abuse within the prior two years.
2. A clinically significant disorder involving the allergy, cardiovascular, respiratory, renal, gastrointestinal/hepatic, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the clinical investigator).
3. History of allergic response(s) to acetaminophen, mannitol, sucralose or related drugs.
4. History of clinically significant allergies including drug allergies or allergic bronchial asthma.
5. Evidence of chronic or acute infectious diseases.
6. Any clinically significant illness or surgery during the one month prior to Period I (or Period III or Period V) dosing (as determined by the clinical investigator).
7. Taking any drug known to induce or inhibit hepatic drug metabolism within one month prior to the beginning of the study.
8. Receiving any investigational drug within one month prior to Period I (or Period III or Period V) dosing.
9. Taking any prescription medication or any nonprescription medication within two weeks prior to Period I (or Period III or Period V) doing.
10. Donating greater than 150 ml of blood within two months prior to Period I (or Period III or Period V) dosing or donating plasma (e.g. plasmapheresis) within two weeks prior to Period I (or Period III or Period V) dosing.
11. Consumption of caffeine, xanthine-containing products (i.e. coffee, tea, caffeine-containing sodas, colas and chocolate, etc.) and/or alcohol within 48 hours prior to days on which dosing is scheduled and during the periods when blood samples are being collected.
12. Any other medical reason as determined by the clinical investigator.
13. Subject is pregnant or breastfeeding.
14. Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline of ALT peak level within study periods | Blood samples were collected on days 2-7 (before dosing)
  ALT peak level in blood after administration

SECONDARY OUTCOMES:
- Incidence of peak ALT elevations > 1X ULN within study periods; | Day 1-7
  The blood concentration of ALT.
- Incidence of peak ALT elevations > 2X ULN within study periods; | Day 1-7
  The blood concentration of ALT.
- Incidence of peak ALT elevations > 3X ULN within study periods; | Day 1-7
  The blood concentration of ALT.
- Incidence of peak ALT elevations > 5X ULN within study periods; | Day 1-7
  The blood concentration of ALT.
- Incidence of peak ALT elevations > 8X ULN within study periods; | Day 1-7
  The blood concentration of ALT.
- Incidence of total bilirubin ≥ 2.5mg/dL within study periods; | Day 1-7
  The blood concentration of total bilirubin.
- Hepatic failure rate (hepatic encephalopathy, ascites, total bilirubin ≥ 2.5mg/dL or liver transplantation) within study periods; | Day 1-7
  The blood concentration of hepatic encephalopathy, ascites, total bilirubin.
- The time-interval weighted area under the curve (AUC) of free plasma acetaminophen-cysteine (AAP-Cys) and AAP-Cys adducts within study periods. | Day 1-7
  The blood concentration of free plasma acetaminophen-cysteine (AAP-Cys) and AAP-Cys adducts
- The time-interval weighted area under the curve (AUC) of ALT level within study periods | Day 1-7
  The blood concentration of ALT.

OTHER OUTCOMES:
- Incidence of adverse events | Day 1-12
  Safety
- Clinical laboratory test | Day 1-12
  Concentrations of acetaminophen in plasma
- Clinical laboratory test | Day 1-12
  Concentrations of acetaminophen metabolites (AAP-Glc) in plasma
- Clinical laboratory test | Day 1-12
  Concentrations of acetaminophen metabolites (AAP-Sul) in plasma
- Clinical laboratory test | Day 1-12
  Concentrations of acetaminophen metabolites (GS-AAP) in plasma
- Clinical laboratory test | Day 1-12
  Concentrations of acetaminophen metabolites (AAP-Cys) in plasma
- Clinical laboratory test | Day 1-12
  Concentrations of acetaminophen metabolites (AAP-NAC) in plasma
- Vital sign | Day 1-12
  Heart rate (bpm)
- Vital sign | Day 1-12
  Blood pressure (mmHg)
- Vital sign | Day 1-12
  Temperature (℃)

CONTACTS AND LOCATIONS:
Overall Officials: TeYu Mr Lin, Dr., Principal Investigator — Principal Investigator
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu District, Taiwan